CLINICAL TRIAL: NCT07062471
Title: Prospective, Multi-center, Single-arm Study of the Shockwave Medical SkyRunner Carotid Intravascular Lithotripsy (IVL) System for the Treatment of Calcified Carotid Arteries Prior to Trans-Carotid Stenting (SKYWARD Trans-Carotid IDE Study)
Brief Title: Study of the Shockwave Medical SkyRunner Carotid Intravascular Lithotripsy (IVL) System for the Treatment of Calcified Carotid Arteries Prior to Trans-Carotid Stenting (SKYWARD Trans-Carotid IDE [Investigational Device Exemption] Study)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry); Yale Cardiovascular Research Group (Other); Cardiovascular Research Foundation, New York (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 75489
Record Dates: First submitted 2025-06-30; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Carotid Artery Calcification; Carotid Artery Diseases
Keywords: IVL; Carotid Calcification; Calcification
MeSH Terms: conditions — Carotid Artery Diseases; Calcinosis

STUDY DESIGN:
Intervention Model Description: The objective of the study is to assess the safety and effectiveness of IVL [Intravascular Lithotripsy] to treat calcified carotid arteries prior to stenting with commercially available trans-carotid stent systems in patients at high risk for complications from CEA (carotid endarterectomy).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Calcified Carotid Artery (Experimental): Up to 160 subjects with calcified carotid arteries to be treated with intravascular lithotripsy (IVL) prior to stenting with commercially available trans-carotid stent systems in patients at high risk for complications from carotid endarterectomy (CEA) will be enrolled in the study.
  Interventions: Device: Carotid Intravascular Lithotripsy (IVL)

INTERVENTIONS:
Device: Carotid Intravascular Lithotripsy (IVL) — The Shockwave Medical Intravascular Lithotripsy (IVL) System with the Shockwave SkyRunner Carotid IVL Catheter is intended for lithotripsy- enhanced balloon dilatation of ≥ 3 mm thick calcified lesions in the carotid arteries prior to stenting. Not for use for treating massive exophytic (mushroom-like) or irregular endoluminal carotid calcification, or in the coronary or cerebral arteries.
  Other Names: Intravascular Lithotripsy (IVL)

SUMMARY:
Prospective, Multi-center, Single-arm Study of the Shockwave Medical SkyRunner Carotid Intravascular Lithotripsy (IVL) System for the Treatment of Calcified Carotid Arteries prior to Trans-Carotid Stenting (SKYWARD Trans-Carotid IDE Study)

DETAILED DESCRIPTION:
To assess the safety and effectiveness of the Shockwave Medical SkyRunner Carotid IVL System for the treatment of calcified carotid arteries prior to stenting with commercially available trans-carotid stent systems in patients at high risk for complications from carotid endarterectomy (CEA).

Up to 160 subjects will be enrolled at up to 25 sites in the United States (US). The estimated study duration is approximately 40 months. Study subjects will be followed through discharge, 30 days, 6, 12, and 24 months.

ELIGIBILITY:
General Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient is able and willing to comply with all assessments in the study.
3. Patient has been informed of the nature of the study, agrees to participate and has signed the approved informed consent form.
4. Patient approved for inclusion by a Patient Screening Committee.
5. Patient must have a life expectancy > 1 year at the time of the index procedure with no planned major cardiac intervention or surgery within 30 days following the index procedure.

   Angiographic Inclusion Criteria:
6. Patient has a discrete lesion located in the internal carotid artery (ICA) with or without involvement of the carotid bifurcation.
7. Target lesion must meet all requirements for commercially available trans-carotid stent systems (refer to IFU for requirements) and investigator intends to treat the target lesion with a single stent.
8. Patient must meet one of the following criteria regarding neurological symptom status and degree of stenosis by duplex ultrasound in combination with CT or MR angiography:

   1. Symptomatic: ≥ 50% stenosis of the internal carotid artery and the patient has a history of stroke, TIA and/or amaurosis fugax within 180 days of the procedure ipsilateral to the carotid artery to be treated.

      OR
   2. Asymptomatic: ≥ 70% stenosis of the internal carotid artery without any neurological symptoms.
9. Patient has evidence of circumferential calcification of the stenotic lesion defined as ≥ 3 mm thickness of calcification as determined by Computed Tomography Angiography (CTA).
10. Patient is high risk for CEA defined as meeting at least one anatomic or clinical high-risk condition listed below:

Anatomic High Risk Inclusion Criteria:

* Contralateral Carotid artery occlusion.
* Tandem Stenoses > 70%.
* High cervical carotid artery stenosis.
* Restenosis after carotid endarterectomy.
* Bilateral carotid artery stenosis requiring treatment within 30 days after index treatment.
* Hostile neck anatomy but which the Investigator deems safe for trans- carotid access including but not limited to:

  * Prior neck irradiation
  * Radical neck dissection
  * Cervical spine immobility

Clinical High Risk Inclusion Criteria:

* Patient is ≥ 70 years of age.
* Patient has congestive heart failure (CHF) - New York Heart Association (NYHA) Functional Class III or IV.
* Patient has severe pulmonary disease (COPD) with either FEV < 50% predicted or chronic oxygen therapy or resting PO2 of < 60 mmHg (room air).
* Patient has a history of angina Canadian Cardiovascular Society (CCS) class 3 or 4 or unstable angina.
* Patient has known severe left ventricular dysfunction LVEF < 30%.
* Patient had a myocardial infarction > 72 hours and < 6 weeks prior to procedure.
* Coronary artery disease with two or more vessels with ≥ 70% stenosis.
* Planned coronary artery bypass grafting (CABG) or valve replacement surgery between 31 and 60 days after index procedure.
* Patient has permanent contralateral cranial nerve injury/paralysis.
* Patient has chronic renal insufficiency (serum creatinine ≥ 2.5 mg/dL). Note that patients on dialysis are excluded from study consideration per exclusionary criterion #16.
* Planned abdominal aortic aneurysm repair or peripheral vascular surgery between 31 to 60 days after index procedure.

General Exclusion Criteria:

1. Patient has alternative source of cerebral embolus, including but not limited to:

   1. a history of chronic atrial flutter or atrial fibrillation, or paroxysmal atrial flutter or atrial fibrillation requiring chronic anticoagulation
   2. knowledge of cardiac sources of emboli (e.g., left ventricular aneurysm, intracardiac filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, hemodynamically significant aortic stenosis, endocarditis, mitral stenosis, or left atrial myxoma)
   3. recently (< 60 days) replaced/repaired heart valve (either surgically or percutaneously).
2. Patient has a history of spontaneous intracranial hemorrhage within the past 12 months, a hemorrhagic transformation of an ischemic stroke within the past 60 days or has had a recent stroke (< 7 days) of sufficient size (on CT or MRI) to place the patient at risk of hemorrhagic conversion during the procedure.
3. Patient with a history of major stroke with substantial neurological deficit (NIHSS ≥ 5 or mRS ≥ 3) within 1 month of index procedure.
4. Patient has had a TIA, or amaurosis fugax within 48 hours prior to the procedure.
5. Patient has neurologic illnesses within the past 2 years characterized by fleeting or fixed neurologic or cognitive deficit which cannot be distinguished from TIA or stroke.
6. Patient has an intracranial tumor.
7. Patient has an isolated hemisphere.
8. Patient has an open stoma in the neck.
9. Patient has an unresolved/uncorrected bleeding disorder.
10. Patient had a myocardial infarction (MI) within last 72 hours prior to index procedure.
11. Patient has contralateral laryngeal, lateral recurrent, or vagus nerve injury.
12. Patient has history of intolerance or allergic reaction to contrast material that cannot be adequately premedicated or to any of the required study medications (i.e., antiplatelet agents, statins) or device materials (refer to IFUs).
13. Female patients who are pregnant, nursing, or may become pregnant.
14. Patient is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached its primary endpoint.
15. Patient has other medical, social, or psychological problems that, in the opinion of the investigator, would present difficulty in complying with protocol requirements.
16. Patient is on renal replacement therapy (i.e., dialysis).

    Angiographic Exclusion Criteria:
17. Presence of a previously placed intravascular stent in the target vessel or ipsilateral CCA.
18. A significant CCA inflow or distal/intracranial lesion.
19. Occlusion (TICI 0) or "string sign" > 1 cm of the ipsilateral common or internal carotid artery.
20. An intraluminal filling defect consistent with thrombus.
21. CCA disease that would preclude the use of TCAR per IFU.
22. Presence of extensive or diffuse atherosclerotic disease involving the aortic arch or proximal common carotid artery that would preclude the safe introduction of the study device.
23. Patient has < 5 cm of distance between the clavicle and bifurcation, as assessed by duplex ultrasound.
24. Cerebral aneurysm, symptomatic or > 5 mm or AVM (arteriovenous malformation) of the cerebral vasculature.
25. Massive exophytic (mushroom-like) or irregular endoluminal calcification seen on CTA or fluoroscopy.
26. Failure to successfully cross the guidewire across the target lesion; successful crossing defined as tip of the guidewire distal to the target lesion in the absence of flow-limiting dissections or perforations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint with death, stroke, and myocardial infarction (MI) [Safety] | 30 days
  A composite endpoint with death, stroke (fatal/disabling or non-disabling based on NeuroARC [Neurologic Academic Research Consortium] definitions) and myocardial infarction (MI) (using the SCAI [Society for Cardiovascular Angiography & Intervention] definition for peri- procedural MI and the 4th Universal Definition for spontaneous MI beyond 48 hours) at 30 days post procedure.

SECONDARY OUTCOMES:
Incidence of any stroke | 30 days, 6 months, 12 months, and 24 months
  Incidence of any stroke through 30 days, 6, 12 and 24 months of follow-up, categorized as:
  * Fatal/Disabling or Non-disabling
  * Ipsilateral or Contralateral
  * Hemorrhagic, Ischemic, or Unknown
Proportion of subjects with Device Success without serious angiographic complications | Day 0
  Proportion of subjects with Device Success, defined as the ability of the IVL catheter to fully cross the target lesion and delivery of lithotripsy without serious angiographic complications, defined as severe dissection (Grade D to F), perforation, abrupt closure, or distal embolization on final angiography, as assessed by the core lab.
Proportion of subjects with residual diameter stenosis ≤ 50% | Day 0
  Proportion of subjects with stent delivery with a residual diameter stenosis ≤ 50% (core lab assessed) on final angiography.
Proportion of lesions with a residual stenosis of ≤ 30% | Day 0
  Proportion of lesions with stent delivery with a residual stenosis of ≤ 30% (core lab assessed) on final angiography.
Incidence of Myocardial Infarction (MI) | Day 0, 30 days, 6, 12, and 24 months post procedure
  Incidence of Myocardial Infarction (MI) (using the SCAI definition for peri- procedural MI; using the 4th Universal Definition for spontaneous MI beyond 48 hours) at discharge, 30 days, 6, 12, and 24 months.
Incidence of Transient Ischemic Attack (TIA) | Day 0, 30 days, 6, 12, and 24 months post procedure
  Incidence of Transient Ischemic Attack (TIA) at discharge, 30 days, 6, 12, and 24 months.
Number of patients with change in NIH Stroke Scale | Day 0, 30 days, 6, 12, and 24 months post procedure
  Change in NIH [National Institutes of Health] Stroke Scale (NIHSS) at post-treatment (within 24 hours), discharge, 30 days, 6, 12 and 24 months.
Cranial Nerve Palsy Assessment for Cranial nerve injury | Day 0, 30 days, 6, 12, and 24 months post procedure
  Cranial Nerve Palsy Assessment for cranial nerve injury at discharge, 30 days, 6, 12 and 24 months.
Neurological function assessed by Modified Rankin Scale (mRS) | Day 0, 30 days, 6, 12, and 24 months post procedure
  Neurological function assessed by Modified Rankin Scale at discharge, 30 days, 6, 12 and 24 months.
  Grade 0 - No symptoms Grade 1 - No significant disability despite symptoms Grade 2 - Slight Disability Grade 3 - Moderate Disability Grade 4 - Moderately Severe Disability Grade 5 - Severe Disability Grade 6 - Deceased
Incidence of all cause death | 30 days, 6, 12, and 24 months post procedure
  Incidence of all cause death, at 30 days, 6, 12 and 24 months.
Number of participants with Clinically-Driven target lesion revascularization (CD-TLR) | Day 0, 30 days, 6, 12, and 24 months post procedure
  Incidence of Clinically-driven target lesion revascularization (CD-TLR), adjudicated by the CEC, at discharge, 30 days, 6, 12 and 24 months.
Number of participants with in-stent restenosis as assessed by DUS core lab | 6, 12, and 24 months post procedure
  Incidence of In-stent restenosis (defined as > 70% restenosis per Duplex Ultrasound (DUS), assessed by DUS core lab, at 6, 12, and 24 months.

IPD SHARING:
Plan to Share IPD: No